CLINICAL TRIAL: NCT07154264
Title: A Phase 2 Study of DZD8586 Combination Therapy in Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: A Study of DZD8586 Combination in CLL/SLL (TAI-SHAN10)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dizal (Jiangsu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dizal Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2025B0001
Record Dates: First submitted 2025-08-18; First posted 2025-09-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of DZD8586 and Venetoclax (Experimental): DZD8586 will be taken orally once daily on days 1-28 of each cycle. Venetoclax will be taken orally once daily on days 1-28 starting from cycle 4 day 1.
  Interventions: Drug: DZD8586; Drug: Venetoclax

INTERVENTIONS:
Drug: DZD8586 — DZD8586 will be taken orally once daily on days 1-28 of each cycle.
  Other Names: Birelentinib
Drug: Venetoclax — Venetoclax will be taken orally once daily on days 1-28 starting from cycle 4 day 1.

SUMMARY:
This is a phase 2 study to investigate the efficacy and safety of DZD8586 in combination in participants with CLL/SLL.

This study consists of two parts: Part A is the safety lead-in phase, and Part B is the dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years of age.
2. ECOG performance status 0-2, and life expectancy ≥ 6 months.
3. Confirmed newly diagnosis or treatment naïve CLL/SLL with indication for treatment.
4. Patients with SLL must have at least one measurable lesion.
5. Adequate bone marrow reserve and organ functions.
6. Willing to comply with contraceptive restrictions.

Exclusion Criteria:

1. Any of previous or current treatment prohibited by protocol.
2. Any unresolved > grade 1 drug-related adverse events.
3. Known or suspected Richter's transformation, or prolymphocytic leukemia.
4. CNS involvement.
5. Active infection.
6. Any of severe cardiac or pulmonary abnormalities.
7. Poorly controlled autoimmune anemia or autoimmune thrombocytopenia.
8. Poorly controlled gastrointestinal disorder, inadequate absorption of medication or other systemic diseases.
9. Prior malignancy within the past 3 years.
10. Known allergy to study drugs, any of the ingredients of the study drugs, or xanthine oxidase inhibitors or rasburicase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of Adverse Events | 30 days after the last dose
Part B: 2-year progression free survival (PFS) rate assessed by investigator | Approximately 5 years

SECONDARY OUTCOMES:
Part A: PFS assessed by investigator | Approximately 5 years
Part A: Objective response rate (ORR) assessed by investigator | Approximately 5 years
Part B: ORR assessed by investigator | Approximately 5 years
Part B: Incidence of Adverse Events | 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Niu, Principal Investigator — West China Hospital
Locations (15):
- China (15):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No